CLINICAL TRIAL: NCT05111132
Title: Can Peripheral NIRS Predict the Response to a Fluid Challenge in Pediatric Patients: An Interventional Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Lulia Scolobiuc, Principal investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: P2021/055/CCB B4062021000019
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 7.5 ml/kg (Experimental): Group 1, receiving a fluid challenge of 7,5 ml/kg in 5 minutes
  Interventions: Diagnostic Test: Fluid challenge (cristalloïd, NaCl 0,9%)
- 12.5 ml/kg (Experimental): Group 2, 12.5 ml/kg of fluid challenge in 5 minutes
  Interventions: Diagnostic Test: Fluid challenge (cristalloïd, NaCl 0,9%)

INTERVENTIONS:
Diagnostic Test: Fluid challenge (cristalloïd, NaCl 0,9%) — A fluid challenge according to group will be administrated by infusion pump

SUMMARY:
This study will be conducted on pediatric patients up to 14 years of age. The effect of two fluid challenge regimes on cerebral and peripheral NIRS will be assessed, in a randomized double blinded controlled trial. The findings will be correlated with two ultrasound measures, previously validated as markers of fluid responsiveness.

DETAILED DESCRIPTION:
The patients will be recruited during the preoperative consultation. After inhalational induction and placement of all monitors, an intravenous access is established. After induction and securing of the airway via endotracheal tube or laryngeal mask, we note the reference values of all parameters. A pre-fluid challenge ultrasound is done, to assess the inferior vena cava distensibillity index, and the Vmax aortic peak flow velocity. After this the fluid challenge is performed. The second ultrasound measures are done after the fluid challenge. Finally an ultrasound is performed at the end of the operation, before emergence, to assess wether the standard peroperative fluid therapy has affecter these measures. NIBP, SpO2, HR, RR, NIRS values will be noted throughout the whole perioperative period. THe end-goald is to correlate the ultrasound findings to the NIRS-values, and see wether the NIRS can be used as a monitor of fluid therapy in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* all operations excepting cardiac surgery
* BMI < 30
* ages 1-14 years

Exclusion Criteria:

* any cardiac affection (congenital unoperated heart disease, arrythmias)
* icterus
* refusal

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Effect of fluid challenge on quadricipital NIRS | 6 hours
  We will assess the effect of fluid challenge on muscular quadricipital in correlation with validated parameters for fluid therapy (dynamic parameters measured by ultrasound: IVC distensibility indec, Vmax aorta)
Effect of fluid challenge on deltoid NIRS | 6 hours
  We will assess the effect of fluid challenge on muscular deltoid NIRS in correlation with validated parameters for fluid therapy (dynamic parameters measured by ultrasound: IVC distensibility indec, Vmax aorta)
Effect of fluid challenge on cerebbral NIRS | 6 hours
  We will assess the effect of fluid challenge on cerebral NIRS in correlation with validated parameters for fluid therapy (dynamic parameters measured by ultrasound: IVC distensibility indec, Vmax aorta)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Pandin, MD, Study Director — Medical doctor
Locations (1):
- Erasmus Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No